CLINICAL TRIAL: NCT00537017
Title: A Phase 2, 36-Week, Open-Label, Uncontrolled Safety Follow-up Study Assessing SCH 420814 (Preladenant) 5 mg BID (P05175)
Brief Title: Follow Up Safety Study of SCH 420814 in Subjects With Parkinson's Disease (P05175)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05175; MK-3814-021 (Other: Merck)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Movement Disorders; Brain Diseases
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Movement Disorders; Brain Diseases | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preladenant 5 mg BID (Experimental): Preladenant 5 mg twice daily (BID) given open-label for 36 weeks to participants with moderate to severe Parkinson's Disease who are on a long-term and stable L-dopa treatment regimen.
  Interventions: Drug: Preladenant; Drug: L-dopa; Drug: Other Parkinson's Disease treatments

INTERVENTIONS:
Drug: Preladenant — 5 mg BID capsules
  Other Names: SCH 420814; Privadenant
Drug: L-dopa — Participants must receive L-dopa as part of their usual ongoing treatment for Parkinson's Disease. L-dopa is often administered concomitantly with a dopa decarboxylase inhibitor (e.g., carbidopa).
Drug: Other Parkinson's Disease treatments — Participants may also receive other drugs as part of their usual ongoing treatment for Parkinson's Disease, such as dopamine agonists (e.g., pramipexole) and/or the catechol-O methyl transferase (COMT) inhibitor entacapone.

SUMMARY:
The purpose of this study is to assess the long term safety of SCH 420814 (preladenant) in participants with moderate to severe Parkinson's Disease who are taking an L-Dopa/dopa decarboxylase inhibitor and/or dopamine agonist. All participants must have participated in the main study (P04501; NCT00406029) entitled "A Phase 2, 12 Week, Double Blind, Dose Finding, Placebo Controlled Study to Assess the Efficacy and Safety of a Range of SCH 420814 Doses in Subjects With Moderate to Severe Parkinson's Disease Experiencing Motor Fluctuations and Dyskinesias."

ELIGIBILITY:
Inclusion Criteria:

* Participants must have participated in P04501.
* Participants must be >=30 years of age, with a diagnosis of moderate to severe idiopathic Parkinson's disease.
* Participants must have been on a regimen of L-Dopa and/or a dopamine agonist.

Exclusion Criteria:

* Participants who discontinued from Study P04501 because they experienced a serious adverse event (SAE)
* Participants with any form of drug-induced or atypical parkinsonism, cognitive impairment, or psychosis
* Participants taking tolcapone
* Participants who are participating in any other clinical study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-11-23 (Actual); Primary Completion 2009-11-19 (Actual); Study Completion 2009-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Factor SA, Wolski K, Togasaki DM, Huyck S, Cantillon M, Ho TW, Hauser RA, Pourcher E. Long-term safety and efficacy of preladenant in subjects with fluctuating Parkinson's disease. Mov Disord. 2013 Jun;28(6):817-20. doi: 10.1002/mds.25395. Epub 2013 Apr 15. PMID 23589371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from Study P04501 (NCT00406029) were enrolled into this study (Treatment Phase [TP] and Follow-up Phase [FUP]).
Pre-assignment Details: Screening for entry into the TP was performed over an 8 day period.
Groups:
- Preladenant 5 mg BID: Preladenant 5 mg BID given open-label for 36 weeks to participants with moderate to severe Parkinson's Disease who are on a long-term and stable L-dopa treatment regimen.
Period: Treatment Phase
Arm/Group | Preladenant 5 mg BID
Started | 140
Completed | 106
Not Completed | 34
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 2
Period: Follow-up Phase
Arm/Group | Preladenant 5 mg BID
Started | 135 (All TP participants were eligible for FUP entry. 5 participants completing TP did not enter FUP.)
Completed | 126
Not Completed | 9
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 95

OUTCOME MEASURES:

1. Secondary Outcome: Time Spent in "Off" State Per Day
Description: Participant diaires recorded time spent in the "off" state at half-hourly intervals for at least 3 full days before scheduled visits. "Off" time is defined as when the participant's medication is not working as subjectively determined by the participant and his/her physician. Higher "off" time values relative to Baseline (BL) signify that the Parkinson's disease symptoms are worse (i.e., participant can only move slowly or not at all). BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
Hours/day
  P04501 BL (n=133) | 5.6 (2.1)
  P04501 BL_LA (n=133) | 4.3 (3.0)
  Week 4 (n=132) | 4.2 (2.8)
  Week 8 (n=119) | 4.0 (3.0)
  Week 12 (n=119) | 3.7 (2.8)
  Week 24 (n=110) | 3.7 (3.0)
  Week 36 (n=99) | 4.1 (3.3)
  Endpoint (n=133) | 4.2 (3.3)

2. Secondary Outcome: Awake Time Per Day in the "on" State
Description: Participant diaries recorded time spent in the "on" state at half-hourly intervals for at least 3 full days before scheduled visits. "On" time is defined as when the participant's medication is working as subjectively determined by the participant and his/her physician. Higher "on" time values relative to BL mean that the Parkinson's disease symptoms are better or absent (i.e., participant can move well). BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 10.6 (2.1)
  P04501 BL (Last Assessment) (n=133) | 11.7 (3.2)
  Week 4 (n=132) | 11.9 (2.9)
  Week 8 (n=119) | 12.0 (3.0)
  Week 12 (n=119) | 12.1 (3.2)
  Week 24 (n=110) | 12.2 (3.4)
  Week 36 (n=99) | 11.9 (3.5)
  Endpoint (n=133) | 11.8 (3.4)

3. Secondary Outcome: Time Spent in the "on" State With no Dyskinesias
Description: Participant diaries recorded time spent in the "on" state with no dyskinesias at half-hourly intervals for at least 3 full days before scheduled visits. "On" time is defined as when the participant's medication is working as subjectively determined by the participant and his/her physician. Dyskinesias are a side effect of long-term therapy with L-dopa consisting of unintentional twisting and/or turning movements that occur in the "on" time. Higher values relative to BL signify an improvement in the Parkinson's disease symptoms (i.e., participant can move well) concomitant with no dyskinesias. BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 6.3 (3.2)
  P04501 BL_LA (n=133) | 7.1 (4.4)
  Week 4 (n=132) | 6.8 (4.1)
  Week 8 (n=119) | 6.9 (3.9)
  Week 12 (n=119) | 7.0 (4.3)
  Week 24 (n=110) | 6.9 (4.4)
  Week 36 (n=99) | 6.9 (4.4)
  Endpoint (n=133) | 6.6 (4.3)

4. Secondary Outcome: Time Spent in the "on" State With Troublesome Dyskinesias
Description: Participant diaries recorded time spent in the "on" state with troublesome dyskinesias at half-hourly intervals for at least 3 full days before scheduled visits. "On" time is defined as when the participant's medication is working as subjectively determined by the participant and his/her physician. Dyskinesias are a side effect of long-term therapy with L-dopa consisting of unintentional twisting and/or turning movements that occur in the "on" time; troublesome dyskinesias interfere with function or cause discomfort. Higher values relative to BL signify that the Parkinson's disease symptoms are better or absent (i.e., participant can move well) concomitant with troublesome dyskinesias. BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 1.0 (1.6)
  P04501 BL_LA (n=133) | 1.2 (2.1)
  Week 4 (n=132) | 1.4 (2.4)
  Week 8 (n=119) | 1.3 (1.9)
  Week 12 (n=119) | 1.3 (2.1)
  Week 24 (n=110) | 1.4 (2.4)
  Week 36 (n=99) | 1.4 (2.4)
  Endpoint (n=133) | 1.5 (2.4)

5. Secondary Outcome: Time Spent in the "on" State Without Troublesome Dyskinesia
Description: Participant diaries recorded time spent in the "on" state without troublesome dyskinesias at half-hourly intervals for at least 3 full days before scheduled visits. "On" time is defined as when the participant's medication is working as subjectively determined by the participant and his/her physician. Dyskinesias are a side effect of long-term therapy with L-dopa consisting of unintentional twisting and/or turning movements that occur in the "on" time; troublesome dyskinesias interfere with function or cause discomfort. Higher values relative to BL signify that the Parkinson's disease symptoms are better or absent (i.e., participant can move well) concomitant with absence of troublesome dyskinesias. BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 3.3 (2.8)
  P04501 BL_LA (n=133) | 3.4 (3.4)
  Week 4 (n=132) | 3.7 (3.5)
  Week 8 (n=119) | 3.8 (3.7)
  Week 12 (n=119) | 3.8 (3.9)
  Week 24 (n=110) | 3.8 (3.7)
  Week 36 (n=99) | 3.6 (3.7)
  Endpoint (n=133) | 3.8 (3.6)

6. Secondary Outcome: Absolute Duration of Dyskinesias
Description: Participant diaries recorded time spent in the "on" state with dyskinesias at half-hourly intervals for at least 3 full days before scheduled visits. "On" time is defined as when the participant's medication is working as subjectively determined by the participant and his/her physician. Dyskinesias are a side effect of long-term therapy with L-dopa consisting of unintentional twisting and/or turning movements that occur in the "on" time. Higher values relative to BL signify worsening of dyskinesia (i.e., more time spent with dyskinesia). BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 4.3 (3.5)
  P04501 BL_LA (n=133) | 4.6 (4.3)
  Week 4 (n=132) | 5.1 (4.5)
  Week 8 (n=119) | 5.1 (4.5)
  Week 12 (n=119) | 5.2 (4.6)
  Week 24 (n=110) | 5.2 (4.6)
  Week 36 (n=99) | 5.0 (4.5)
  Endpoint (n=133) | 5.3 (4.5)

7. Secondary Outcome: Total Sleep Time
Description: Participant diaries recorded time spent in the sleep state at half-hourly intervals for at least 3 full days before scheduled visits. BL was determined using two methods: 1) P04501 BL refers to the starting BL of the double-blind base study P04501 and 2) P04501 BL_LA refers to BL as defined by the last assessment taken in P04501. Endpoint refers to the last observed result for participants within P05175.
Time Frame: Baseline (P04501 BL; P04501 BL_LA), Week 4, Week 8, Week 12, Week 24, Week 36
Population: All participants with a baseline value and at least one post-baseline value were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
hours/day
  P04501 BL (n=133) | 7.6 (1.6)
  P04501 BL_LA (n=133) | 7.8 (1.7)
  Week 4 (n=132) | 7.7 (1.6)
  Week 8 (n=119) | 7.8 (1.7)
  Week 12 (n=119) | 7.8 (1.7)
  Week 24 (n=110) | 7.7 (1.9)
  Week 36 (n=99) | 7.9 (1.7)
  Endpoint (n=133) | 7.8 (1.6)

8. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure. A serious adverse event is an adverse event that that results in death, life threatening adverse event, permanent or significant disability / unfitness for work, hospital treatment (i.e., admission to hospital) or prolongation of a patient's length of stay, or congenital deformity or birth defect.
Time Frame: Up to 42 weeks
Population: All participants who received treatment with study drug were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Preladenant 5 mg BID
Number analyzed (Participants) | 140
Participants | 123

ADVERSE EVENTS:
Time Frame: Up to 42 weeks
Description: All participants who received treatment with study drug were included in the analysis.
Arm/Group | Preladenant 5 mg BID
Serious Adverse Events (participants affected / at risk) | 22/140
Other Adverse Events (participants affected / at risk) | 96/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 5 mg BID (N=140)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Amaurosis Fugax (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Abasia (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2)
Completed Suicide (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (2)
Hallucination, Visual (Psychiatric disorders) | 1 (1)
Hallucinations, Mixed (Psychiatric disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Benign Tumour Excision (Surgical and medical procedures) | 1 (1)
Inguinal Hernia Repair (Surgical and medical procedures) | 1 (1)
Shoulder Arthroplasty (Surgical and medical procedures) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 5 mg BID (N=140)
Constipation (Gastrointestinal disorders) | 25 (26)
Diarrhoea (Gastrointestinal disorders) | 11 (14)
Nausea (Gastrointestinal disorders) | 9 (10)
Influenza (Infections and infestations) | 9 (11)
Nasopharyngitis (Infections and infestations) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 17 (28)
Blood Creatine Phosphokinase Increased (Investigations) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15)
Back Pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 (10)
Dyskinesia (Nervous system disorders) | 46 (63)
Headache (Nervous system disorders) | 13 (17)
Parkinson's Disease (Nervous system disorders) | 18 (23)
Somnolence (Nervous system disorders) | 15 (16)
Insomnia (Psychiatric disorders) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.